CLINICAL TRIAL: NCT06912256
Title: Influence Of Individualized Two Weeks Mild Sleep Restriction On Tactical Performance During Small-Sided Games In National Male Under-19 Football Players: A Randomized Trial
Brief Title: The Effects of Individualised Short-term Sleep Restriction on Tactical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: José Afonso Coelho Neves (Other)
Responsible Party: Sponsor-Investigator, José Afonso Coelho Neves, Supervisor of the lead author's Master Thesis, Universidade do Porto
Organization: Universidade do Porto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CEFADE 9 2023
Record Dates: First submitted 2025-03-23; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Sleep Restriction
Keywords: sleep restriction; performance; tactical; small-sided games; soccer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep restriction (Experimental): During the intervention period (i.e., 9 consecutive days), the intervention group started the sleep protocol, sleeping only the quantity of hours defined for their individual chronic partial sleep restriction (15% of usual daily sleep hours). The amount and quality of sleep obtained were daily monitored through actigraphy devices, and all the players filled in a sleep diary when they woke up. During this period, players performed the SSGs in two different moments (moment 1 and moment 2), interspersed by 4 days.
  Interventions: Behavioral: Sleep restriction
- Controls (No Intervention): Same intervention (i.e., soccer training and tests) as the other arm, but with no sleep restriction.

INTERVENTIONS:
Behavioral: Sleep restriction — During the intervention period (i.e., 9 consecutive days), the intervention group started the sleep protocol, sleeping only the quantity of hours defined for their individual chronic partial sleep restriction (15% of the usual sleep time). The amount and quality of sleep obtained were daily monitored through actigraphy devices, and all the players filled in a sleep diary when they woke up. During this period, players performed the SSGs in two different moments (moment 1 and moment 2), interspersed by 4 days.
  Arms: Sleep restriction

SUMMARY:
The goal was to evaluate the influence that chronic sleep restriction may have on football players tactical performance during small-sided games. By using a relative sleep restriction (i.e., by reducing the normal sleep duration by 15%) instead of an absolute sleep restriction (e.g., 3-4 hours), different sleep schedules were applied, according to the players individual sleep profile. It was hypothesized that the player's performance would be impaired, particularly their tactical behaviors when performing a 4x4 small-sided game format.

DETAILED DESCRIPTION:
An impairment on cognitive and physical performance is commonly suggested in literature. However, there is a lack of information regarding sport-specific parameters. Thus, the present study aimed to examine whether chronic sleep restriction during 9 consecutive days impairs the tactical performance of football players during small-sided games (SSGs). A total of sixteen national level male football players wore wrist actigraphy units during night sleep throughout the study. Players were randomized into two groups: intervention (IG), and control (CG). The first four days corresponded to a familiarization period, where players were informed about the study procedures and started using wrist actigraphy. Throughout the next seven consecutive days, the characterization phase of sleep players profile (i.e., baseline) was collected and analyzed. Then, players entered the intervention phase, where the IG slept 15% less than routine. During this 9-days period, players performed a 4x4 SSGs in two moments (moment 1 and moment 2) with a week interval. The SSGs were recorded using a video camera and subsequently analyzed using the Game Performance Assessment Instrument.

ELIGIBILITY:
Inclusion Criteria:

* Soccer players classified as Tier 3, corresponding to the National Level in accordance to McKay et al. (2022), as they represented the under-19 team playing in the Portuguese National Championship 1st Division.

Exclusion Criteria:

* 1) players with previously identified sleep disorders;
* 2) players with injuries that prevented them from playing SSGs.

Max Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Game Performance Assessment Instrument (GPAI) | Applied once in week 1 and once again in week 2
  According to study purposes, tactical performance was defined as the main variables. Tactical analysis was performed using the Game Performance Assessment Instrument (GPAI), a tool designed to evaluate the individual tactical behavior (Memmert & Harvey, 2008; Oslin, Mitchell, & Griffin, 1998). It consists of seven components, two of which are evaluated when the player has the ball and the remaining five when the player does not have the ball possession. For example, decisions made about what to do with the ball during the game, and motor skill execution were classified as appropriate/efficient or inappropriate/inefficient. The main index proposed by Oslin et al. (1998) was calculated: Game Performance (GP). Based on actions deemed appropriate or inappropriate, the final score can range from 0 to 100%, with higher values denoting better outcomes.

SECONDARY OUTCOMES:
Sleep efficiency | Collected daily during the two weeks of the intervention
  The objective sleep data was collected using three axial accelerometers (ActiGraph LLC wGT3X-BT, Pensacola, USA) placed on the non-dominant wrist. To analyze the wrist actigraphy data, the ActiLife LLC Pro software (v6.13.3, Pensacola, USA) was used with a sampling frequency of 50Hz and an epoch of activity counts of 60s. Sleep efficiency (SE, percentage of time in bed that was spent asleep; CV=7%) was determined using the Sadeh's algorithm.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport, University of Porto, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No
Sensitive data belonging to a club, so we only had permission to report the statistical treatment, but not sharing the IPD.